CLINICAL TRIAL: NCT00941330
Title: Randomized Phase II Trial of Pre-Operative Docetaxel-Cytoxan (TC) or Exemestane in Patients With Hormone Receptor-Positive Breast Cancers With Recurrence Scores Greater Than 10 (≥ 11) and Less Than 25 (≤ 24)
Brief Title: Exemestane or Docetaxel-Cytoxan in Low Recurrence Score Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Elisavet Paplomata, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012969; WCI1534-08 (Other: Other)
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Breast, Male; Breast, Female
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Exemestane (Experimental): ARM A: Patients will be treated with exemestane.
  Interventions: Drug: Exemestane
- B: Docetaxel and Cytoxan (Active Comparator): ARM B: Patients will be treated with docetaxel and cytoxan.
  Interventions: Drug: Docetaxel; Drug: Cytoxan

INTERVENTIONS:
Drug: Exemestane — 25 mg daily by mouth for 6 to 12 months.
  Other Names: Aromasin
  Arms: A: Exemestane
Drug: Docetaxel — Docetaxel (75 mg/m²) into a vein once every 3 weeks for 6 cycles (6 times in about 24 weeks).
  Other Names: Taxotere
  Arms: B: Docetaxel and Cytoxan
Drug: Cytoxan — Cytoxan (600 mg/m²) into a vein once every 3 weeks for 6 cycles (6 times in about 24 weeks).
  Other Names: Cyclophosphamide
  Arms: B: Docetaxel and Cytoxan

SUMMARY:
The patients are being asked to take part in this study because they have a hormone receptor-positive breast cancer (contains estrogen and/or progesterone receptors) and their doctor has told them that they have an option to receive chemotherapy or hormonal therapy before surgery. The purpose of this study is to assess if chemotherapy using docetaxel and cytoxan (TC) or hormonal therapy using exemestane can shrink the size of their breast tumor and allow them to preserve the breast or have less extensive surgery on their breast.

DETAILED DESCRIPTION:
The purpose of this study is to assess if chemotherapy using docetaxel and cytoxan (TC) or hormonal therapy using exemestane can shrink the size of your breast tumor and allow you to preserve your breast or have less extensive surgery on your breast. Additionally, by receiving chemotherapy or hormonal therapy before surgery, we will be able to determine if the treatment you receive is effective in treating your cancer. Prior to entering this study, a special test, called the Oncotype DX assay, will be performed on a small amount of your cancer from the biopsy you had at the time you were diagnosed with breast cancer, to determine the likelihood that your cancer will benefit from and shrink with chemotherapy and hormonal therapy. You will only be eligible to enter this study if the recurrence score of your cancer determined using the Oncotype DX assay is less than or equal to 24. Patients with hormone receptor-positive breast cancers with recurrence scores less than or equal to 24 have been previously demonstrated to obtain a larger benefit from hormonal therapy, compared to chemotherapy, when these agents are given after surgery. The ability of hormonal agents and chemotherapy to shrink cancers prior to surgery has not been specifically examined in hormone receptor-positive cancers with recurrence scores less than or equal to 24.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Histologically or cytologically confirmed breast carcinoma.
* Early stage breast cancer (T1c-3, clinically node-negative-3 [cN0-3], CM0).
* Pre-treatment biopsy with the following characteristics:

  * Hormone receptor-positive cancer as defined as ER and/or progesterone receptor (PR)-positive by standard immunohistochemistry (IHC)
  * HER2-negative (HER2 ≤ 2 by IHC; if HER2 2+ by IHC must be fluorescent in situ hybridization [FISH] non-amplified)
  * Recurrence score < 25 using Oncotype DX 21-gene recurrence score assay
* Patients must have measurable disease as defined by palpable lesion with both diameters ≥ 1 cm measurable with caliper or a positive mammogram or ultrasound with at least one dimension ≥ 1 cm. Screening mammogram of the contralateral breast must be performed within past 12 months per standard practice guidelines. Clip placement is required for study entry.
* Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within 14 days of study enrollment if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a diagnostic mammogram of the affected breast or MRI must be done within 2 months prior to study enrollment, defined as date of signed, informed consent. If clinically indicated, staging xrays and scans must be done within 28 days of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Adequate organ function within 14 days of study entry:

  * Bone marrow function: absolute neutrophil count (ANC) ≥ 1500/mm³, Hgb > 8.0 g/dl and platelet count ≥ 100,000/mm³.
  * Hepatic function: total bilirubin < upper limit of normal (ULN). Serum glutamic oxaloacetic transaminase (SGOT) (AST) or serum glutamic pyruvic transaminase (SGPT) (ALT) and alkaline phosphatase ≤ 1.5 x ULN).
  * Renal function: calculated creatinine clearance (CrCl) ≥ 30 mL/min using the Cockcroft Gault equation.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Evidence of disease outside the breast or chest wall, except ipsilateral axillary or internal mammary lymph nodes.
* Prior chemotherapy, hormonal therapy, biologic therapy or radiation therapy for breast cancer.
* Pregnant or lactating women are not eligible. Women of childbearing potential must have a negative serum pregnancy test completed within 7 days of study entry, and use an appropriate form of birth control throughout the trial period.
* Medical, psychological or surgical condition which the investigator feels might compromise study participation.
* Patients with history within the last 5 years of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies who remain disease free for greater than five years are eligible.
* Evidence of peripheral or sensory neuropathy.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 are excluded from participation.
* Serious, uncontrolled, concurrent infection(s).
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months prior to study entry.
* Major surgery within 28 days of study entry.
* Evidence of central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisavet Paplomata, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2009 to December 2014, patients were recruited at Winship Cancer Institute of Emory University, Emory University Hospital Midtown, and Grady Health System, all in Atlanta, Georgia.
Pre-assignment Details: Five patients were not assigned to a treatment arm. One patient was ineligible for the study due to a low Oncotype score. Three patients did not like randomized treatment. One patient had disease progression.
Period: Overall Study
Arm/Group | A: Exemestane | B: Docetaxel and Cytoxan
Started | 15 | 11
Completed | 14 | 9
Not Completed | 1 | 2
Not completed — Other | 1 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Exemestane | B: Docetaxel and Cytoxan | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: Patients must have measurable disease by clinical examination.
  Pathologic complete response (pCR): Absence of invasive breast cancer in the breast (mastectomy or lumpectomy) specimen at the time of definitive surgery. Presence of in situ cancer alone will be considered a pCR but may be recorded separately.
  If pathologic stage was the same as clinical stage, it was called stable; if it was higher, upstaged (worse outcome); if lower, downstaged (better outcome). Pathologic stage was determined by Emory board-certified pathologists.
Time Frame: At time of definitive surgery
Population: One patient in Arm B did not have surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Exemestane | B: Docetaxel and Cytoxan
Number analyzed (Participants) | 14 | 8
Participants
  Downstaged | 5 | 1
  Stable | 4 | 2
  Upstaged | 5 | 5

2. Secondary Outcome: Response Rate by Imaging
Description: Arm A and recurrence score ≤10: Patients will have radiologic assessment of response to exemestane by clinical examination every 4 weeks and by radiologic assessment every 2 months. Once maximal response has been achieved (stable disease for 2 months after at least 4 months of treatment by radiologic assessment) or when 12 months of therapy has been given patients will proceed to surgery.
  Arm B: Patients will be assessed for surgery after 6 cycles of docetaxel and cytoxan (TC) (18 weeks).
  On arm A and recurrence score ≤10 patients will be reassessed for surgery once maximal radiologic response is achieved.
  On arm B, patients will be reassessed for surgery after 6 cycles of TC (18 weeks).
  Radiographic images were analyzed by a breast radiologist who looked at preoperative and postoperative breast mass imaging. If mass was smaller/less extensive, it was considered improved.
Time Frame: Every 2 months up to 3 years
Population: Data were not available for 5 patients (4 withdrew and 1 did not have surgery).
Measure: Count of Participants; unit: Participants
Arm/Group | A: Exemestane | B: Docetaxel and Cytoxan
Number analyzed (Participants) | 15 | 6
Participants
  Improved | 9 | 2
  Stable | 6 | 4

ADVERSE EVENTS:
Arm/Group | A: Exemestane | B: Docetaxel and Cytoxan
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/11
Other Adverse Events (participants affected / at risk) | 13/15 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Exemestane (N=15) | B: Docetaxel and Cytoxan (N=11)
Gastroenteritis and Severe Diarrhea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Exemestane (N=15) | B: Docetaxel and Cytoxan (N=11)
Fever (General disorders) | 1 | 1
Elevated Liver Enzymes (Hepatobiliary disorders) | 0 | 1
Lower Extremity Edema (General disorders) | 1 | 2
Fatigue (General disorders) | 7 | 9
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Bloating (General disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hot Flashes (General disorders) | 8 | 2
Headache (General disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Nausea (General disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dry Mouth (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Dizziness (General disorders) | 1 | 1
Hypokalemia (Blood and lymphatic system disorders) | 1 | 0
Gait Disturbance (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Oral Mucositis (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Floaters (Eye disorders) | 1 | 0
Bruising (Blood and lymphatic system disorders) | 2 | 0
Depression (Psychiatric disorders) | 4 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2
Insomnia (General disorders) | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Memory Impairment (Nervous system disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chest Pain (General disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Allergic Reaction (Immune system disorders) | 0 | 2
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Dysgeusia (General disorders) | 0 | 1
Watery Eyes (Eye disorders) | 0 | 1
Weight Gain (Metabolism and nutrition disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Irritability (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes